CLINICAL TRIAL: NCT01318642
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of AMG 479 or Placebo in Combination With Gemcitabine as First-line Therapy for Locally Advanced Unresectable Adenocarcinoma of the Pancreas
Brief Title: Ganitumab in Locally Advanced Unresectable Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NCT01318642: Planned independent DMC Interim review: ended for futility
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080261; 2010-023978-39 (EudraCT Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-05

CONDITIONS: Adenocarcinoma of the Pancreas; Locally Advanced; Unresectable
Keywords: Adenocarcinoma; pancreas; pancreatic cancer; local; unresectable; stage II; stage III
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Gemcitabine; ganitumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + Gemcitabine (Active Comparator): Arm 2: AMG479-placebo IV days 1 and 15 plus gemcitabine 1000mg/m2 IV days 1, 8, and 15 of a 28 day cycle
  Interventions: Drug: Gemcitabine; Drug: Placebo
- AMG 479 20 mg/kg + Gemcitabine (Experimental): ARM 1: AMG 479 20mg/kg IV days 1 and 15 plus gemcitabine 1000mg/m2 IV days 1, 8, and 15 of a 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: AMG 479

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine on days 1, 8, and 15, followed by placebo on days 1 and 15 of every 28 day cycle.
  Other Names: Gemzar
Drug: AMG 479 — Gemcitabine on days 1, 8, and 15, followed by AMG 479 20 mg/kg on days 1 and 15 of every 28 day cycle.
  Other Names: gemcitabine = Gemzar
  Arms: AMG 479 20 mg/kg + Gemcitabine
Drug: Placebo — Gemcitabine on Days 1, 8, and 15 followed by Placebo 20 mg/kg on days 1 and 15 of every 28 day cycle
  Arms: Placebo + Gemcitabine

SUMMARY:
This study is a phase 2, multicenter, randomized, double-blind, active placebo-controlled trial of AMG 479 or placebo in combination with gemcitabine as first-line therapy for locally advanced unresectable adenocarinoma of the pancreas. Approximately 150 subjects will be randomized in a 1:1 ratio to AMG 479 and gemcitabine, or gemcitabine and placebo. Randomization will be stratified by ECOG (0 or 1).

Gemcitabine will be given on days 1, 8, and 15, followed by AMG 479 on days 1 and 15 of every 28 day cycle. Treatment will continue until radiographic disease progression, unacceptable toxicity, withdrawal of consent, or start of a new anti-cancer therapy.

DETAILED DESCRIPTION:
This study is a phase 2, multicenter, randomized, double-blind, active placebo-controlled trial of AMG 479 or placebo in combination with gemcitabine as first-line therapy for locally advanced unresectable adenocarinoma of the pancreas. Approximately 150 subjects will be randomized in a 1:1 ratio to AMG 479 and gemcitabine, or gemcitabine and placebo. Randomization will be stratified by ECOG (0 or 1).

Gemcitabine will be given on days 1, 8, and 15, followed by AMG 479 on days 1 and 15 of every 28 day cycle. Treatment will continue until radiographic disease progression, unacceptable toxicity, withdrawal of consent, or start of a new anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed locally advanced adenocarcinoma of the pancreas that is unresectable, per institutional practice
* Radiologically measurable and/or non-measurable disease as defined by RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Men or women >/= 18 years of age
* Adequate organ function

Exclusion Criteria:

* Early (stage I) or metastatic (stage IV) disease
* Islet cell, acinar cell carcinoma, non-adenocarcinoma, (eg, lymphoma, sarcoma, etc), adenocarcinoma originating from biliary tree or cystadenocarcinoma
* External biliary drain
* Currently treated or previously treated with biologic, small molecule, immunotherapy, chemotherapy (ie, including gemcitabine), or other agents for pancreatic cancer
* Currently treated or previously treated with radiotherapy, or chemoradiotherapy for pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2012-11-27 (Actual); Study Completion 2012-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (2):
  - Research Site, San Francisco, California
  - Research Site, Knoxville, Tennessee
- Austria (3):
  - Research Site, Salzburg
  - Research Site, Steyr
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Edegem
  - Research Site, La Louvière
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Herlev, Denmark
- Research Site, Hamburg, Germany
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Szolnok
- Poland (3):
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Russia (4):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Madrid
- United Kingdom (3):
  - Guys Hospital, London
  - Research Site, London
  - Research Site, Preston

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4804122/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Safety Population was used for all summaries (including serious and non-serious adverse events). Only 8/10 subjects received at least 1 dose of protocol-specified treatment and therefore were included in the Safety Population.
Period: Overall Study
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Started | 5 | 3
Completed (Completed defined as receiving at least one dose of study drug.) | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (11.8) | 63.0 (8.7) | 68.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Subjects with locally advanced unresectable adenocarcinoma of the pancreas [Count of Participants; unit: Participants] | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is Progression-free Survival (PFS) as Defined as the Time From Randomization to Progression (Per RECIST v1.1) or Death.
Description: The time from randomization to progression (per RECIST version 1.1) or death from any cause. Disease progression per RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From randomization to the date of either disease progression or death, up to 181 days progression or death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Months | NA [NA to NA] — lack of participants with events | NA [NA to NA] — lack of participants with events

2. Secondary Outcome: Overall Survival
Description: OS - time from study day 1 to death (by any cause)
Time Frame: Up to 181 days
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Months | NA [NA to NA] — lack of participants with events | NA [NA to NA] — lack of participants with events

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Measured via CTCAE v3.0
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Participants | 5 | 3

4. Secondary Outcome: Progression Free Survival Rate and Overall Survival Rate at at 3 and 6 Months, Objective Response Rate, Disease Control Rate
Description: PFS rates - subjects with disease progression (PD) or death at the timepoint; OS rates - subjects alive at the timepoint; ORR - tumor response assessment of either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST); DCR - subjects with PR, CR, or SD Per RECIST: CR=disappearance of all target lesions; PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Disease progression=at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study; stable disease is disease that is not partial or progressed
Time Frame: Up to 181 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Participants
  Progression Free Survival Rate at 3 months | 2 | 0
  Progression Free Survival Rate at 6 months | 2 | 0
  Overall Survival Rate at 3 months | 5 | 3
  Overall Survival Rate at 6 months | 4 | 3
  Objective Response Rate | NA — lack of participants with events (e.g. PR, CR) | NA — lack of participants with events (e.g. PR, CR)
  Disease Control Rate | NA — lack of participants with events (e.g. PR, CR, SD) | NA — lack of participants with events (e.g. PR, CR, SD)

5. Secondary Outcome: Duration of Response
Description: DOR - time from the first observation of an objective response (subjects with CR or PR) to the time of PD or death; Per RECIST: CR=disappearance of all target lesions; PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Disease progression=at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study; stable disease is disease that is not partial or progressed
Time Frame: Up to 181 days
Measure: Mean (Full Range); unit: Months
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Months | NA [NA to NA] — lack of participants with events (eg CR or PR) | NA [NA to NA] — lack of participants with events (eg CR or PR)

6. Secondary Outcome: Number of Participants With Anti-AMG 479 Antibodies
Description: post-dose anti-AMG 479 antibody positive rate
Time Frame: Up to 181 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For Adverse Events: from randomization through 30 (+3) days after the last administration of protocol specified therapy, up to 4 months. For Mortality: from randomization to the end of the study, up to 187 days.
Arm/Group | Placebo + Gemcitabine | AMG 479 20 mg/kg + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=5) | AMG 479 20 mg/kg + Gemcitabine (N=3)
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=5) | AMG 479 20 mg/kg + Gemcitabine (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Fatigue (General disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early. Only the safety data is provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes